CLINICAL TRIAL: NCT03967457
Title: Comprehensive Study on the Quality of Life in Cervical Cancer Patients: A Prospective Cohort Study
Brief Title: Comprehensive Study on the Quality of Life in Cervical Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: CCQOL
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Quality of Life; Cervical Cancer; Urodynamics; Rectum Dynamics; Sex Dysfunction; Pelvic Floor Disorders; Ovarian Reserve Function; Survivorship; Disease-free Survival; Overall Survival
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples for the testing of ovarian reserve function
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: questionnaires survey — Including four kinds of questionnaires: European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 (V3); EORTC QLQ-CX24; Eligibility Criteria (FSFI); and Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFIQ-7)
Diagnostic Test: Urodynamic testing — Urodynamic testing consists of important urodynamic parameters including:
  Bladder capacity at the first void sense Bladder capacity at normal desire to void Bladder capacity at strong desire to void Qmax Qave Pves at Qmax Pdet at Qmax Cves at SDV Cdet at SDV Residual urine volume
Diagnostic Test: Rectum dynamics testing — Rectum dynamics testing consists of important parameters of rectum activities
Diagnostic Test: ovarian reserve function — Testing for ovarian reserve function consists of:
  Follicle-stimulating hormone Estradiol Anti-mullerian hormone Inhibin B

SUMMARY:
This is prospective cohort study. All the patients with primary cervical cancer in the future three years in Peking Union Medical College Hospital will be included in this study. Before and after the major therapy (including at least radical hysterectomy and/or radiotherapy), the patients accept (1) the questionnaires survey about quality of life; (2) urodynamic testing; (3) rectum dynamics testing and (4) ovarian reserve function. The survival outcomes (disease-free survival and overall survival) will be supplemented as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Primary uterine cervical carcinomas
* Aged 18 or older
* Accepting major therapy (including at least radical hysterectomy and/or radiotherapy) in the study center
* Informed consents delivered

Exclusion Criteria:

* Not meeting any of the inclusion criteria
* Not accepting any of the four kinds of evaluations for quality of life
* Recurrent patients
* Not achieving response after above major therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with primary cervical cancer in the future three years in Peking Union Medical College Hospital will be included in this study. They should be 18 years or older, accepting major therapy (including at least radical hysterectomy and/or radiotherapy) in the study cente and achieving response after the major therapy.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Scores from EORTC QLQ-C30 | Change from the baseline of four weeks before major therapy at following-up. The standard scores ranges from 0 to 100, and the higher score, the more inferior quality of life.
  Scores calculated from European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30
Scores from EORTC QLQ-CX24 | Change from the baseline of four weeks before major therapy at following-up. The standard scores ranges from 0 to 100, and the higher score, the more inferior quality of life.
  Scores calculated from EORTC QLQ-CX24

SECONDARY OUTCOMES:
Concentration of follicle-stimulating hormone | Change from the baseline of four weeks before major therapy at following-up
  Follicle-stimulating hormone tested in peripheral blood
Concentration of estradiol | Change from the baseline of four weeks before major therapy at following-up
  Estradiol tested in peripheral blood
Concentration of anti-mullerian hormone | Change from the baseline of four weeks before major therapy at following-up
  Anti-mullerian hormone tested in peripheral blood
Concentration of inhibin B | Change from the baseline of four weeks before major therapy at following-up
  Inhibin B tested in peripheral blood
Bladder capacity at the first void sense | Change from the baseline of four weeks before major therapy at following-up
  Bladder capacity at the first void sense tested by urodynamic testing
Bladder capacity at normal desire to void | Change from the baseline of four weeks before major therapy at following-up
  Bladder capacity at normal desire to void tested by urodynamic testing
Bladder capacity at strong desire to void | Change from the baseline of four weeks before major therapy at following-up
  Bladder capacity at strong desire to void tested by urodynamic testing
Maximun flow rate | Change from the baseline of four weeks before major therapy at following-up
  Maximun flow rate tested by urodynamic testing
Average flow rate | Change from the baseline of four weeks before major therapy at following-up
  Average flow rate tested by urodynamic testing
Bladder pressure at maximun flow rate | Change from the baseline of four weeks before major therapy at following-up
  Bladder pressure at maximun flow rate tested by urodynamic testing
Detrusor pressure at maximun flow rate | Change from the baseline of four weeks before major therapy at following-up
  Detrusor pressure at maximun flow rate tested by urodynamic testing
Bladder compliance at strong desire to void | Change from the baseline of four weeks before major therapy at following-up
  Bladder compliance at strong desire to void tested by urodynamic testing
Detrusor compliance at strong desire to void | Change from the baseline of four weeks before major therapy at following-up
  Detrusor compliance at strong desire to void tested by urodynamic testing
Residual urine volume | Change from the baseline of four weeks before major therapy at following-up
  Residual urine volume tested by urodynamic testing
Anal sphincter pressure | Change from the baseline of four weeks before major therapy at following-up
  Anal sphincter pressure tested by rectum dynamic testing

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No